CLINICAL TRIAL: NCT01811017
Title: Clinical Evaluation of 755nm Alexandrite Laser Versus Nanosecond 755nm Alexandrite
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN12-PICO_MGH_TB
Record Dates: First submitted 2012-12-06; First posted 2013-03-14 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Tattoos
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 755nm Alexandrite Laser (Experimental): 755nm Alexandrite Laser
  Interventions: Device: 755nm Alexandrite Laser
- Nanosecond 755nm Alexandrite Laser (Experimental): Nanosecond 755nm Alexandrite Laser
  Interventions: Device: 755nm Alexandrite Laser

INTERVENTIONS:
Device: 755nm Alexandrite Laser — 755nm Alexandrite Laser

SUMMARY:
Compare the efficacy of the 755nm Alexandrite laser to the nanosecond 755nm Alexandrite laser for the removal of unwanted tattoos using photographic evaluation and histological findings.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 85 years old?
2. Has unwanted non-cosmetic tattoo(s) and wishes to undergo laser treatments
3. Is willing to consent to participate in the study.
4. Is willing to shield the tattoo completely from sun exposure
5. Signs informed consent form
6. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits.

Exclusion Criteria:

1. Subjects who are unwilling to consent to tattoos
2. Subjects mentally ill or incompetent
3. Subjects is unwilling to have photographs taken and used in publications or scientific presentations
4. Subjects who are prisoners
5. Subjects with recent sun exposure and suntan in the area to be treated
6. Allergic tattoos (hypersensitivity to tattoo ink)
7. History of vitiligo or keloidal scarring
8. Tattoos located on the neck or face including cosmetic tattoos
9. Subjects unwilling to tolerate partial removal of the tattoo in this study
10. Infection or skin disease in the area to be treated
11. Subjects who are immunosuppressed (e.g. HIV)
12. Subject is pregnant or nursing
13. Use of oral isotretinoin within past 12 months
14. History of squamous cell carcinoma or melanoma
15. Is allergic to Lidocaine, tetracaine or Xylocaine with epinephrine.
16. Has any other reason determined by the physician to be ineligible to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Photographic Evaluation of Tattoo Clearance | up to 3 months post last treatment

SECONDARY OUTCOMES:
Subject biopsy sampling | up to 3 months post last treatment
  Histological evaluation of tissue samples pre-treatment and post-treatment

OTHER OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | up to 3 months post last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Boston Va Medical Center, Boston, Massachusetts, United States